CLINICAL TRIAL: NCT07022431
Title: Effects of a Strength Training Program With High Cognitive Engagement on Health, Physical Condition, and Quality of Life in People With Alzheimer's Disease
Brief Title: Effects of a Cognitive-Engaging Strength Training Program on Health, Physical Condition, and Quality of Life in People With Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Alejandro Muñoz López, Assistant Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SICEIA-2024-001871
Record Dates: First submitted 2024-07-26; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Cognitive Function; High Cognitive Demand Exercises; Strength Training
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strength training (Experimental): Participants will perform a cognitively demanding exercise while simultaneously performing strength training. With each repetition, the software will display in numbers the average concentric power output performed by the participants. Based on the benefits of performing a cognitively demanding physical exercise, participants will be asked to repeat out loud the value of the average concentric power output of the previous repetition while performing the next one.
  Interventions: Other: Interval strength training
- Control group (No Intervention): These patients only receive the usual treatment for their pathology.

INTERVENTIONS:
Other: Interval strength training — The intervention involves interval strength training with biofeedback and real-time decision-making for Alzheimer's patients. Participants will complete 24 sessions, each including a circuit of strength exercises using rotational inertial devices (flywheels). Exercises, such as leg press, seated row, and bicep curl, will be randomly ordered, with load progression based on performance stability. Each session includes five sets per exercise, performed in a circuit, with a total of 15 sets over approximately 45 minutes. Real-time monitoring using a rotary encoder will track effort, and participants will continue each set until a 30% drop in average power is detected, ensuring consistent relative effort across sets.
  Additionally, participants will engage in cognitively demanding tasks during training by verbally reporting the average power of the previous repetition while performing the next one. This dual-task approach aims to maximize both physical and cognitive engagement.
  Arms: Strength training

SUMMARY:
The primary objective of this project is to examine the impact of a strength training program with high cognitive demands on cognitive function, motor skills, physical fitness, and quality of life in individuals with Alzheimer's disease and mild cognitive impairment. This randomized controlled trial will involve participants for a total of five months. Initial two weeks will be for cognitive, physical fitness, quality of life, and specific biochemical profile evaluations, along with familiarization sessions with the exercise routine. The experimental group will then undertake a supervised strength training program twice a week for 16 weeks. The final two weeks will involve re-evaluations of all initial assessments. Participants will be randomized into a control group and an intervention group with a minimum of 17 individuals each. Stratification criteria for randomization include physical activity level, number of Alzheimer's disease-related risk factors, extent of brain damage based on MRI biomarkers, and clinical dementia rating scores.

DETAILED DESCRIPTION:
Objectives and Hypotheses:

The main objective of this project is to study the effects of a physical exercise program based on strength training with high cognitive implications on cognitive, motor, conditional function, and quality of life in people with Alzheimer's Disease with mild cognitive impairment.

Design:

This study follows a randomized controlled experimental design. Participants will be involved in the study for a total of five months. During the first two weeks, participants will be evaluated regarding their cognitive function, physical condition, quality of life, and specific biochemical profile. Additionally, during these two weeks, they will undergo familiarization sessions with the exercise routine. Subsequently, the experimental group will perform supervised strength training, two days a week with 48-72 hours of separation between sessions, for a total of 16 weeks. The last two weeks will involve retesting all the evaluations conducted during screening and pre-intervention.

Participants will be stratified and randomized into a control group (minimum n=17) and an intervention group (minimum n=17). Randomization will consider the following strata: 1) level of physical activity, 2) number of risk factors associated with Alzheimer's disease, 3) degree of brain damage according to MRI neuroimaging biomarkers, and 4) Clinical Dementia Rating (CDR). The level of physical activity will have two groups: 1) physically active, those engaging in moderate to vigorous activity for more than 150 minutes per week, or 2) physically inactive (less than 150 minutes per week), evaluated through the adapted International Physical Activity Questionnaire for the elderly (IPAQ-E). The number of associated risk factors will have the following groups: 1) presents 3 or fewer factors, 2) presents between 4 and 7 factors, 3) presents 8 or more factors. The degree of brain damage according to biomarkers will have the following groups, based on hippocampal atrophy degree by volume: 1) 30th percentile of participants, 2) 30th to 60th percentile, 3) 60th percentile onwards. The CDR score will have the following groups: 1) up to questionable dementia (CDR < 0.5), 2) from mild dementia (CDR > 1). The control group will be instructed to maintain their normal life habits concerning physical activity levels, cognitive training, and diet. The experimental group will follow the training plan described later. The design of this study follows the procedures previously approved in the Declaration of Helsinki - ethical principles for medical research involving human subjects.

Participants:

The research will be announced to obtain participants through the following channels: 1) advertisements in the local press, 2) mass email to potential participants, 3) Alzheimer's, memory, and/or dementia associations, 4) medical specialists. The screening process will follow this strategy:

Telephone interview: potential candidates living in Seville city or nearby metropolitan area.

In-person interview: a cognitive assessment will be conducted with a specific neuropsychological battery to help define the patient's neuropsychological profile. First, a screening test will be conducted, and if the patient meets the inclusion criteria, the standardized cognitive assessment will be completed with other cognitive tests.

Medical evaluation: a complete clinical history will be conducted, including pre-assessment of possible hidden risks contraindicated for physical activity, carried out by a sports medicine specialist. Additionally, resting blood pressure will be evaluated.

After the cognitive assessment, we will obtain a list of possible study participants. Since we require a total of 34 people for the necessary statistical power, we will conduct the study with a total of 50 people, due to possible exclusions that may occur in the medical evaluation, according to the established exclusion criteria.

To safeguard confidentiality and anonymity, the following measures will be implemented:

Informed consent: Before participating, subjects will be informed about the use of their data and must give their explicit consent to participate in the study.

Data coding: Unique codes will be assigned to participants instead of using their real names in all records and documents, thus maintaining their anonymity (e.g., "RTP1" according to the order in the sample). This task will be carried out by the data management researcher GRP.

Secure storage: Collected data will be securely stored on secure servers, with access restricted only to authorized personnel (GRP), to prevent unauthorized disclosures. The storage location will be Microsoft's OneDrive, protected by a two-factor code for access in addition to a personal password.

Limited disclosure: Only the information necessary for the study purposes will be shared, avoiding the disclosure of personal details.

Publications and presentations: In any publication or presentation related to the study, only aggregated or anonymous data will be used to protect participants' identities.

Sample size:

This study will require a total sample size of 34 participants. This is the minimum required sample size according to calculations performed to achieve a minimum statistical power of 80%: RANOVA test with between-group and within-group interactions, effect size of f= 0.25 (equivalent to a partial eta squared - moderate effect size of 0.06 points), Alpha error probability type I of 0.05, with 2 between-group factors (control and experimental) and 2 within-group factors (pre and post intervention), with a correlation value of 0.5 between repeated measures, and assuming sphericity correction in the used test.

Inclusion and exclusion criteria for participants:

The inclusion criteria will be: 1) being between 65 and 75 years old, 2) any gender, 3) meeting the criteria for early-stage AD dementia (GDS 4) (according to DSM-IV-TR and NINCDS-ADRDA criteria), 4) having a score between 15 and 20 on the Mini-Mental State Examination (Trivedi, 2017), indicating moderate cognitive impairment, 5) maintaining a stable pharmacological regimen for at least 30 days before, 6) giving consent to be evaluated through the cognitive screening tests described in this report, 7) availability to attend weekly training sessions in Seville city.

The exclusion criteria will be: 1) presence of heart disease or other conditions contraindicating physical activity, 2) presence of psychiatric disorders, 3) having any musculoskeletal pathology or disorder preventing the proposed exercises or conditional evaluations, 4) having a resting heart rate below 50 or above 100 beats per minute, and 5) having a diagnosed intellectual disability.

For this research project, the following materials will be used:

Takei 5401 handheld dynamometer (Takei Kiki Kogyo, Japan). It will allow measurement of handgrip strength in conditional evaluation tests.

Witty photocells (Microgate, Italy). They will allow measurement of displacement time, as well as calculation of displacement speed, in conditional evaluation tests.

SmartCoach rotary encoder (SmartCoach Tech, USA). It will measure mechanical performance during the execution of each strength training exercise. Additionally, it will provide real-time feedback to adjust training load and perform high cognitive demand tasks simultaneously with the exercise (dual-task).

Omron HEM-7120 blood pressure monitor (OMRON Healthcare Inc., Japan). It will allow measurement of blood pressure and resting heart rate before and after each training session.

Lactate Pro 2 LT-1730 lactate meter (Arkray, Kyoto, Japan). It will allow measurement of lactate produced after various training sessions.

Flywheel Kpulley 2 device (Exxentric, Sweden). Essential training device for the execution of the proposed strength training as the main intervention.

Flywheel Kbox Squat device (Exxentric, Sweden). Essential training device for the execution of the proposed strength training as the main intervention.

RBANS and CDR test battery. They will allow measurement of cognitive function.

Data will be primarily described using the mean of each variable. We will use standard deviation and the 95% confidence interval of the mean as descriptive dispersion measures. Before any analysis, we will check if the sample distribution is normal using a Shapiro-Wilk test. The possible changes produced in training, between the experimental and control groups, will be analyzed through a mixed repeated measures ANOVA, with a within-subjects factor (time, pre vs. post) and a between-subjects factor (groups, experimental vs. control). In case of significant differences, a post hoc analysis with Bonferroni correction will be performed. Additionally, effect size (partial eta squared) will be reported. The significance level will be set at p < 0.05 for all tests. Data analysis will be performed with IBM's SPSS statistical package.

Preliminary Results:

This study aims to determine if a training program based on strength exercises with high cognitive implications improves cognitive, motor, conditional function, and quality of life in people with mild cognitive impairment due to Alzheimer's disease. For the different evaluated aspects, an improvement is expected in the group participating in the proposed training program, compared to the control group.

Limitations and future directions Participant recruitment: finding an adequate number of participants meeting the strict inclusion and exclusion criteria may be challenging. The timeframe for recruitment and evaluation might need adjustments to ensure an adequate sample size.

Adherence to the training program: participants' adherence to the training sessions could vary due to personal or health issues, potentially impacting the results. Strategies to enhance adherence and compliance should be considered.

Generalizability of results: the findings might be limited to individuals with similar demographics, health conditions, and geographic locations as the participants. Future studies should aim to include more diverse populations to improve generalizability.

Long-term effects: this study will focus on short-term outcomes (5 months). Long-term effects of the training program on cognitive, motor, and conditional function, and quality of life should be investigated in future research.

Control group activities: although the control group will be instructed to maintain their normal life habits, potential confounding factors related to their activities outside the study may affect the results. Monitoring control group activities more closely might provide more accurate comparisons.

Calendar and Project Plan:

Project Phases and Timeline:

* Phase 1: Preparation and Recruitment (Month 1) Preparation of recruitment materials and study information Recruitment and screening of participants Obtain informed consent
* Phase 2: Initial Assessment (Months 2-3) Conduct cognitive, physical, and biochemical assessments Familiarization sessions with the exercise routine
* Phase 3: Intervention (Months 4-7) Experimental group: Supervised strength training sessions Control group: Maintain normal life habits Ongoing monitoring and support
* Phase 4: Final Assessment (Months 8-9) Retesting all evaluations conducted during screening and pre-intervention
* Phase 5: Data Analysis and Reporting (Months 10-12)

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for early AD dementia (GDS 4) (according to the DSM-IV-TR and NINCDS-ADRDA criteria)
* Have a score between 15 and 20 on the Mini-Mental State Examination scale (Trivedi, 2017), with criteria for moderate cognitive impairment.
* Maintain a stable pharmacological regimen for at least 30 days prior.
* Give consent to be evaluated using the cognitive screening tests described in this report.
* Be available to attend in person weekly at the headquarters where the training will take place in Seville capital.

Exclusion Criteria:

* Presence of heart disease or other diseases that lead to a contraindication in the practice of physical activity.
* Presence of psychiatric illnesses.
* Having some musculoskeletal pathology or alteration that does not allow the performance of the proposed exercises or proposed conditional evaluations.
* Having a resting heart rate less than 50 or greater than 100 beats per minute.
* Having a diagnosed intellectual disability.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Global cognitive performance | Baseline (pre-intervention, week 0) and immediately after intervention (week 16).
  Assessed using the Total Score from the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Clinical Assessment of Dementia | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Global score obtained from the Clinical Dementia Rating Scale (CDR de Hughes).
Isometric knee flexion-extension strength | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Changes in the isometric knee flexion-extension strength will be assessed using the Biodex isokinetic dynamometer.
Number of repetitions in the 30-second Sit-to-Stand test | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Assessed using the 30-second Sit-to-Stand test. The participant is instructed to rise to a full standing position and sit down as many times as possible within 30 seconds without using the arms. The number of repetitions is recorded.
Handgrip strength | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Changes in the handgrip strength (handgrip test) assessed by Takei 5401
10m walking velocity | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Changes in the time taken to cover 10 meters (10m walk test).
Time to complete the Timed Up and Go test (3 meters) | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Changes in the time needed to stand up from a chair, walk 3 meters, turn, return, and sit down (Timed Up and Go test).
Decrement in walking speed during dual-task 10m walk test | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  To assess possible improvements in dual-task exercises, we will use a variant of the previously described 10-meter walk test. The protocol being the same as above, while walking, participants will be instructed to perform the following cognitive tasks: in the first walk, they will receive the instruction "walk at your usual walking speed while naming the months backwards, starting from January"; in the second walk, they will receive the instruction "walk at your usual walking speed while counting backwards from 50". In total, participants will perform three attempts of each verbal instruction. The best time will be taken as the final result. Finally, the decrement in performing this modified test compared to the original will be calculated, using the following formula ((10m dual task - 10m single task)/10m single task X 100).
Health-related quality of life measured by EuroQol-5D (EQ-5D) | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Quality of life will be assessed using the EuroQol-5D questionnaire (EQ-5D), a standardized instrument to measure health-related quality of life across five dimensions. Both patient and caregiver reports will be considered.
Distance walked in the 6-Minute Walk Test (6MWT) | Baseline (week 0) and immediately after the 12-week intervention (week 16)
  Changes in the distance (in meters) covered during the 6-Minute Walk Test (6MWT), a submaximal aerobic capacity test commonly used in elderly and clinical populations.

SECONDARY OUTCOMES:
Blood lactate concentration | During the 12-week intervention period (weeks 1 to 12)
  Capillary blood lactate levels will be measured before and after one of the two weekly training sessions (randomly selected), throughout the 12-week intervention, in participants assigned to the experimental group.